CLINICAL TRIAL: NCT02976168
Title: Intracranial Pressure and Brain Function: Effects of Head Down Tilt Upon Brain Perfusion and Cognitive Performance
Acronym: IPCog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DLR German Aerospace Center (Other)
Collaborators: Forschungszentrum Juelich (Other); University Hospital, Umeå (Other); University of Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IPCog
Record Dates: First submitted 2016-11-18; First posted 2016-11-29 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Intracranial Hypertension
Keywords: Cognitive functioning; Brain tissue oxygenation; cerebral perfusion; head down tilt
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Horizontal (No Intervention): Subjects will be in horizontal supine Position for 21 hours
- -12° head down tilt (Experimental): Subjects will be in 12° head down supine Position for 21 hours
  Interventions: Other: 12° head down tilt

INTERVENTIONS:
Other: 12° head down tilt — supine head down tilt
  Arms: -12° head down tilt

SUMMARY:
The aim of the study is to understand the relationship between intracranial pressure regulation, cerebral tissue oxygenation and cognitive functioning. More specifically, the study tests the hypothesis that head down tilt will increase intracranial pressure (not measured in this study, but demonstrated in previous studies), will induce venous congestion and facial swelling, decrease intracranial tissue oxygenation and hamper brain functioning. The objectives of the study therefore are to assess young healthy people during head-down tilt (HDT), and to assess cognitive brain functioning, cerebral tissue oxygenation (non-invasively), frontal skin thickness, cerebral perfusion and neuronal functioning via event-related potentials.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy male test subjects that are able and declare in writing their willingness to participate in the entire study and successfully passed the psychological and medical screening
* Aged between 18-55 years old with a Body Mass Index (BMI) of 20-28 kg/m2, weight between 65-100 kg, and a height between 158-195 cm
* Demonstrable medical insurance and official certificate of absence of criminal record

Exclusion Criteria:

* Inability to sleep on the back
* Drug, medication or alcohol abuse (regular consumption of more than 20-30 g alcohol/day)
* Smoking within the past 6 months prior to study commencement
* Migraine or other chronic head aches
* Previous psychiatric illness
* Subjects suffering from weak concentration
* History of psychological or central nervous disorders
* Hiatus hernia
* Gastro-oesophageal reflux
* Diabetes mellitus
* Pronounced orthostatic intolerance (< 10 min standing)
* Kidney disorder: deviations from normal values for creatinine in plasma. (Normal value: Creatinine < 1.20 mg/dl)
* Thyroid gland disorder: deviations from normal values for thyroid stimulating Hormone (TSH) in plasma. (Normal range: TSH 0.55-4.80 mUnits/l)
* Anaemia: Hb under normal values (Normal values of Hb for men: 13.5-17.5 g/l)
* Elevated risk of thrombosis
* High likelihood of coagulopathy assessed by a clinical standard questionnaire
* Chronic back complaints
* History of lumbar surgery
* History of lumbar spine trauma
* Motor or sensory deficits as assessed by neurological examination
* Contraindications against MRI
* Imprisoned at the time of the study
* Taking medications that may impair cognitive function, autonomic function or any of the study procedures
* Ophthalmological conditions including glaucoma, retinopathy, severe cataracts, eye trauma or implants
* Any other medical condition that the investigators consider a contraindication to the study procedures that would make it unsafe or confound the measurements.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in cognitive test battery score | Twice at baseline, and 30 minutes and 20 hours after starting the intervention
  The test battery includes sensomotoric speed, psychomotor vigilance, visual analysis of items, abstract thinking and mathematical processing

SECONDARY OUTCOMES:
Change in mid cerebral artery blood flow velocity | Twice at baseline, and 10 minutes and 19 hours after starting the intervention
  Transcranial Doppler measurements
Change in cerebral tissue oxygenation | Twice at baseline, and 10 minutes and 19 hours after starting the intervention
  Near-infrared measurement
Magnetic resonance Imaging: Change in cerebral blood flow | Once at baseline, and 2 and 19 hours after starting the intervention
  Magnetic resonance imaging will be performed in order to gain information about intracranial blood flow.
Magnetic resonance Imaging: Change in resting state functional MRI (fMRI) | Once at baseline, and 2 and 19 hours after starting the intervention
  Magnetic resonance imaging will be performed to assess resting state functional MRI.
Magnetic resonance Imaging: Change in fMRI Response to decision task | Once at baseline, and 2 and 19 hours after starting the intervention
  Magnetic resonance imaging will be performed in order to assess functional MRI during a decision task combing a reaction time test using a visual stimulus.
Change in jugular vein filling | Once at baseline, and 10 minutes and 19 hours after starting the intervention
  Conventional Imaging ultrasound from jugular veins veins will be used to assess vein cross sections
Change in frontal vein filling | Once at baseline, and 10 minutes and 19 hours after starting the intervention
  Conventional Imaging ultrasound from the frontal veins will be used to assess vein cross sections
Change in P-300 | Twice at baseline, and 30 minutes and 20 hours after starting the intervention
  P-300 will be assessed via an EEG electrode during cognitive test battery
Change in sleep effectiveness | over the entire intervention night
  Polysomnographic recordings
Change in total sleep time | from 22:00 until 6:00 in all nights
  Polysomnographic recordings

OTHER OUTCOMES:
Change in frontal skin thickness | Once at baseline, and 10 minutes and 19 hours after starting the intervention
  Conventional Imaging ultrasound will be used to assess Skin thickness at the frontal skull
Change in arterial blood pressure | Twice at baseline, and 10 minutes and 19 hours after starting the intervention
  arterial blood pressure will be assessed non-invasively from a finger artery during transcranial doppler measurements
Change in heart rate | Twice at baseline, and 10 minutes and 19 hours after starting the intervention
  ECG will be recorded during transcranial doppler measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jörn E Rittweger, MD, Principal Investigator — German Aerospace Center
Locations (1):
- DLR German Aerospace Center, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boschert AL, Elmenhorst D, Gauger P, Li Z, Garcia-Gutierrez MT, Gerlach D, Johannes B, Zange J, Bauer A, Rittweger J. Sleep Is Compromised in -12 degrees Head Down Tilt Position. Front Physiol. 2019 Apr 16;10:397. doi: 10.3389/fphys.2019.00397. eCollection 2019. PMID 31040791